CLINICAL TRIAL: NCT04802057
Title: An Open-label, Long-term, Safety and Tolerability Study of SAR445088 in Participants With Cold Agglutinin Disease Previously Treated With SAR445088 or Never Treated With SAR445088
Brief Title: Safety and Tolerability Study in Adults With Cold Agglutinin Disease Previously Treated With SAR445088 or Never Treated With SAR445088
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bioverativ, a Sanofi company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTS16637; U1111-1244-0808 (Registry Identifier: ICTRP); 2023-510210-68 (Registry Identifier: CTIS); 2019-004423-21 (EudraCT Number)
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Autoimmune Haemolytic Anaemia
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- SAR445088 (Experimental): Repeat dose of SAR445088
  Interventions: Drug: SAR445088

INTERVENTIONS:
Drug: SAR445088 — Pharmaceutical form: solution for injection
  Route of administration: IV and SC (Part 1) IV (Part 2)

SUMMARY:
Primary Objective:

To assess the long-term safety and tolerability in patients with cold agglutinin disease (CAD), after multiple doses of SAR445088

Secondary Objective:

To assess, in patients with cold agglutinin disease (CAD), after multiple doses of SAR445088:

* The long-term effect of SAR445088 on complement mediated hemolysis
* The long-term pharmacodynamics (PD) effect of SAR445088 relating to complement inhibition
* The long-term pharmacokinetic (PK) profile of SAR445088
* The long-term immunogenicity of SAR445088

DETAILED DESCRIPTION:
The screening period for this study is up to 6 weeks. The treatment period for this study will continue for 2 years after last participant entered Part 2 (either having switched from Part 1 or as a SAR445088-naïve participant), or until SAR445088 development is discontinued, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult patients ≥18 years of age with CAD who were previously treated with SAR445088 and met criteria the below criteria for entry into Part 1:

  * met the eligibility criteria of a previous study evaluating SAR445088;
  * successfully enrolled and completed dosing in a previous study evaluating SAR445088;
  * successfully completed end of study procedures in a previous study evaluating SAR445088; and
  * per Investigator judgement, had a favorable benefit-to-risk profile after receiving SAR445088.
* OR were never treated with SAR445088 before entering Part 2, and met the below criteria to establish CAD diagnosis:

  * chronic hemolysis;
  * polyspecific direct antiglobulin test (DAT) positive status;
  * monospecific DAT strongly positive for C3d;
  * cold agglutinin [CAg] titer ≥64 at 4°C;
  * IgG DAT ≤1+;
  * hemoglobin level ≤10 g/dL;
  * elevated bilirubin not attributable to liver disease;
* Documented vaccinations against encapsulated bacterial pathogens given within five years of enrollment and at least 14 days prior to dosing (vaccinations have to be initiated at least 14 days prior to dosing and completed before Week 5 of Part 2).
* Contraception (with double contraception methods) for male and female participants; not pregnant or breastfeeding for female participants; no sperm donation for male participants.
* Having given written informed consent prior to undertaking any study-related procedure.

Exclusion Criteria:

* Cold agglutinin syndrome secondary to infection, rheumatologic disease, or known high-grade hematologic malignancy, or known solid organ tumor.
* Clinically relevant infection within 1 month of enrollment.
* Clinical diagnosis of systemic lupus erythematosus (SLE).
* Treatment with anti-CD20 monotherapy within 3 months or anti-CD20 combination therapies within 6 months prior to screening.
* Concurrent treatment with systemic immunosuppressive agents targeting B- or T-cell function and/or cytotoxic agents within 3 months prior to screening. Concurrent treatment with other systemic immunosuppressants within 5.5 half-lives of the drug prior to screening.
* Any specific complement system inhibitor other than SAR445088 (eg, eculizumab) within 3 months prior to screening.
* Concurrent treatment with systemic corticosteroids other than a stable daily dose equivalent to ≤10 mg/day prednisone within 3 months prior to screening.
* History of hypersensitivity to SAR445088 or any of its components.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-03-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAE) | Day 1 or Day 1-IV to end of study, approximately 6 years
  The number of participants experiencing TEAEs will be reported for the overall safety population.

SECONDARY OUTCOMES:
Mean change from baseline in total bilirubin over time | Day 1 or Day 1-IV to end of study, approximately 6 years
  Assessment of total bilirubin
Mean change from baseline in hemoglobin over time | Day 1 or Day 1-IV to end of study, approximately 6 years
  Assessment of hemoglobin
Mean change from baseline in lactate dehydrogenase over time | Day 1 or Day 1-IV to end of study, approximately 6 years
  Assessment of lactate dehydrogenase
Mean change from baseline in reticulocyte count over time | Day 1 or Day 1-IV to end of study, approximately 6 years
  Assessment of reticulocyte count
Complement System Classical Pathway Levels as Measured by WIESLAB Assay | Day 1 or Day 1-IV to Week 48-IV
  Inhibition by SAR445088 of the complement system classical pathway measured by the WIESLAB assay.
Complement System Alternative Pathway Levels as Measured by WIESLAB Assay | Day 1 to Week 24
  Part 1: Effect of SAR445088 on the complement system alternative pathway measured by the WIESLAB assay.
Mean change in CH50 over time | Day 1 or Day 1-IV to end of study, approximately 6 years
  Complement CH50 is a blood test that helps us determine whether protein abnormalities and deficiencies in the complement system are responsible for any increase in autoimmune activity. It will be assessed using complement assays.
Total Complement Factor C4 Levels | Day 1 or Day 1-IV to end of study, approximately 6 years
  Total C4 Levels will be assessed in plasma using complement assays
PK parameter: Cmax | Day 1 or Day 1-IV to Week 48-IV
  Maximum observed concentration (Cmax) of SAR445088 in plasma will be assessed
PK Parameter: AUC | Day 1 or Day 1-IV to Week 48-IV
  Area under the plasma concentration versus time curve calculated using the trapezoidal method at steady state
Number of participants with anti-SAR445088 antibodies | Day 1 or Day 1-IV to end of study, approximately 6 years
  The immunogenicity for SAR445088 will be assessed by summarizing the number of participants with anti-SAR445088 antibodies (ADA)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (5):
- Investigational Site Number : 2760001, Essen, Germany
- Investigational Site Number : 3800001, Milan, Milano, Italy
- Investigational Site Number : 5280001, Amsterdam, Netherlands
- Investigational Site Number : 5780001, Bergen, Norway
- Investigational Site Number : 8260001, London, London, City of, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LTS16637 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25302&tenant=MT_SNY_9011